CLINICAL TRIAL: NCT01723826
Title: A Multicenter, Open-Label, Long-Term Safety Extension of Phase II Studies ABE4869g and ABE4955g in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: A Long-Term Safety Extension of Studies ABE4869g and ABE4955g in Participants With Mild to Moderate Alzheimer's Disease Treated With Crenezumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN28525; 2012-003242-33 (EudraCT Number)
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — crenezumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Crenezumab (Experimental): Participants will receive intravenous infusion of crenezumab every 4 weeks for 144 weeks.
  Interventions: Drug: Crenezumab

INTERVENTIONS:
Drug: Crenezumab — Participants will receive intravenous infusion of crenezumab every 4 weeks for 144 weeks.
  Other Names: RO5490245

SUMMARY:
This Phase II, open-label extension (OLE), multicenter study will evaluate the long-term safety and tolerability of crenezumab in participants with mild to moderate Alzheimer's disease who have participated in and completed the treatment period of the Phase II Study ABE4869g (NCT01343966) or ABE4955g (NCT01397578). Participants who received placebo in Study ABE4869g (NCT01343966) or ABE4955g (NCT01397578) will receive crenezumab. Anticipated time on study treatment is 144 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in Study ABE4869g or ABE4955g and completion of the Week 73 visit
* Adequate visual and auditory acuity, in the investigator's judgment, to allow for neuropsychological testing
* Availability of a person ("caregiver") who can provide information on activities of daily living and behavior in order to complete the study-specific assessments
* Diagnosis of probable Alzheimer's disease according to the National Institute on Neurological and Communication Disease and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria (McKhann et al. 1984)
* Mini-Mental State Examination (MMSE) score of 10 or more at screening (Folstein et al. 1975)
* For male participants with partners with reproductive potential, agreement to use a reliable means of contraception (e.g., condoms) during the study and for at least 8 weeks following the last dose of study drug
* For female participants, a negative pregnancy test at screening

Exclusion Criteria:

* Early treatment and/or study discontinuation prior to completion of the Week 73 visit of Genentech Study ABE4869g or ABE4955g
* Early discontinuation from the treatment schedule of a prior version of Study GN28525 for safety reasons. If treatment discontinuation occurred for safety reasons, participants may not re-start dosing on extended treatment schedules offered in amendments to Study GN28525
* Inability to tolerate Magnetic Resonance Imaging (MRI) procedures or contraindication to MRI
* Female participants with reproductive potential: Female participants must either have undergone documented surgical sterilization or have not experienced menstruation for at least 12 consecutive months
* Severe or unstable medical condition that, in the opinion of the investigator or Sponsor, would interfere with the participant's ability to complete the study assessments or would require the equivalent of institutional or hospital care
* History or presence of clinically evident vascular disease potentially affecting the brain
* History of severe, clinically significant central nervous system trauma
* History or presence of clinically relevant intracranial tumor
* Presence of infections that affect the brain function or history of infections that resulted in neurologic sequelae
* History or presence of systemic autoimmune disorders potentially causing progressive neurologic disease
* History or presence of a neurologic disease other than Alzheimer's disease that may affect cognition
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins
* Evidence of malignancies (except squamous cell cancer or basal cell cancer of the skin), acute infections, renal failure that requires dialysis, or other unstable medical disease not related to Alzheimer's disease that, in the investigator's opinion, would preclude participant's participation. Cancer that is not being actively treated with anti-cancer therapy or radiotherapy as well as cancers which are considered to have low probability of recurrence are allowed
* History or presence of atrial fibrillation that, in the investigator's judgment, poses a risk for future stroke
* Chronic kidney disease of Stage greater than or equal to (>=) 4, according to the National Kidney Foundation Kidney Disease Outcomes Quality Initiative (NKF KDOQI) guidelines for chronic kidney disease (CKD)
* Impaired hepatic function
* Impaired coagulation (activated partial thromboplastin time [aPTT] greater than [>] 1.2 times upper limit of normal [ULN])
* Platelet count less than (<) 100,000 per microliter (mcL)
* Presence at screening of superficial siderosis of central nervous system, more than 8 cerebral microhemorrhages, or evidence of a prior cerebral macrohemorrhage
* Presence at screening of any other significant cerebral abnormalities, including ARIA-E
* Treatment with anticoagulation medications within 2 weeks prior to enrollment. Clopidogrel, dipyridamole, and aspirin are permitted
* Treatment with anticholinergic antidepressants, typical antipsychotics, or barbiturates within 2 weeks prior to enrollment. All other antidepressants and atypical antipsychotics are allowed with certain restrictions as defined in the protocol
* Chronic use of opiates, opioids, or benzodiazepines
* Any biologic therapy within 75 weeks prior to enrollment
* Any investigational agent (other than crenezumab) within 75 weeks prior to enrollment
* Treatment with anticholinergic antidepressants, typical antipsychotics, barbiturates, or narcotics within 5 half-lives or 3 months prior to screening, whichever is longer. All other antidepressants and atypical antipsychotics are allowed. Chronic use of benzodiazepines is not allowed; however, the intermittent use of benzodiazepines is allowed, except within 2 days prior to any neurocognitive assessment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2012-12-07 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (86):
- United States (47):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Banner Sun Health Research Insitute, Sun City, Arizona
  - Pharmacology Research Inst, Encino, California
  - Margolin Brain Institute, Fresno, California
  - Univ of CA San Diego; Neurosciences Comp.Alzheimer's, La Jolla, California
  - USC School of Medicine, Los Angeles, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - Pharmacology Research Inst, Newport Beach, California
  - Pacific Neuroscience Med Grp, Oxnard, California
  - Stanford Univ Medical Center, Palo Alto, California
  - University of California Davis Medical System, Sacramento, California
  - Pacific Research Network - PRN, San Diego, California
  - Uni of California San Francisco, San Francisco, California
  - Redwood Regional Medical Group, Santa Rosa, California
  - Yale University, New Haven, Connecticut
  - Florida Atlantic University; College of Medicine, Boca Raton, Florida
  - Meridien Research, Brooksville, Florida
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Miami Jewish Health Systems; Clinical Research, Miami, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Bioclinica Research, Orlando, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Dekalb Neurology Associates, Decatur, Georgia
  - Rush Alzheimer's Disease Cntr., Chicago, Illinois
  - Alexian Brothers Neurosci Inst, Elk Grove Village, Illinois
  - Indiana Univ School of Med, Indianapolis, Indiana
  - Louisiana Research Associates, New Orleans, Louisiana
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Millennium Psychiatric Associates, LLC, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo; Center for Brain Research, Las Vegas, Nevada
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - NeuroCognitive Institute, Mount Arlington, New Jersey
  - Empire Neurology, PC, Latham, New York
  - Litwin Zucker Research Ctr.; Feinstein Inst. Med. Rsch., Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center; Monroe Community Hospital, Rochester, New York
  - Investigational Drug Service; Univ of Rochester Medical Ctr, Rochester, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Summit Research Network Inc., Portland, Oregon
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Medical Uni of South Carolina, North Charleston, South Carolina
  - Alzheimers Disease & Memory Disorders Center; Department of Neurology Baylor College of Medicine, Houston, Texas
  - Clinical Neuroscience Research Associates, Inc., Bennington, Vermont
- Canada (13):
  - The Med Arts Health Rsrch Grp, Kelowna, British Columbia
  - University of British Columbia Hospital; Division of Neurology, Vancouver, British Columbia
  - Capitol District Health Authority, Halilfax, Nova Scotia
  - Jbn Medical Diagnostic Services Inc., Burlington, Ontario
  - Hotel Dieu Hospital, Kingston, Ontario
  - St. Joseph's HC-Parkwood Hosp, London, Ontario
  - Bruyere Continuing Care, Ottawa, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program (Neurology Research Inc.), Toronto, Ontario
  - Clinique Neuro Rive-Sud, Greenfield Park, Quebec
  - Hôpital Maisonneuve-Rosemont/Polyclinique;Recherche Clinique, Montreal, Quebec
  - CHAUQ Hopital Enfant-Jesus, Québec, Quebec
  - McGill Univeristy; Douglas Mental Health University Institute; Neurological and Psychiatric, Verdun, Quebec
- France (6):
  - Hopital neurologique Pierre Wertheimer - CHU Lyon; Neurologie, Bron
  - CHU de Limoges Hopital Dupuytren; Service de Medecine Geriatrique, Limoges
  - Hopital Central; Neurologie, Nancy
  - Hopital Nord Laennec, Nantes
  - CHU de Rouen Hopital; Service de Neurologie, Rouen
  - Hôpital Civil de Strasbourg, Strasbourg
- Germany (6):
  - Univ Berlin; Klin fur Psychi & Psycho Charite, Berlin
  - Bezirkskrankenhaus Günzburg, Günzburg
  - Zentralinstitut fuer Seelische Gesundheit, Mannheim
  - Ludwig-Maximilians-Univ., München
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Universitätsklinik Tübingen; Psychiatrie und Psychotherapie, Tübingen
- Spain (6):
  - Fundació ACE, BArcelon, Barcelona
  - Hospital General de Catalunya, San Cugat Del Valles, Barcelona
  - Policlinica Guipuzcoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital de Cruces; Servicio de Neurologia, Barakaldo, Vizcaya
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Clinica Ruber, 4 planta; Servicio de Neurologia, Madrid
- United Kingdom (8):
  - The Rice Centre; Royal United Hospital, Bath
  - West London Research Unit; Brentford Lodge, Brentford
  - Royal Sussex County Hospital, CIRU Level 5, Brighton
  - Glasgow Memory Clinic, Glasgow
  - The National Hospital for Neurology & Neurosurgery; Dementia Research Center, London, GT LON
  - Southampton General Hospital; Pharmacy, Southampton
  - Moorgreen Hospital; Memory Assessment & Rsch Ctr, Southampton
  - Great Western Hosp.; Kingshill Research Ctr, Swindon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 360 participants were enrolled at 83 sites across 6 countries.
Pre-assignment Details: Participants who completed either Phase II Study NCT01343966 (ABE4869g) or NCT01397578 (ABE4955g) and had Mini-Mental State Examination (MMSE) score of 10 or more at the time of screening were included. Participant flow is represented based on the safety population by treatment received.
Groups:
- PCP PL - OLE CREN SC - OLE CREN IV: Participants who on their placebo-controlled portion [PCP]/parent study received placebo (PL) and who on this open-label extension (OLE) study initially received crenezumab (CREN) subcutaneously (SC) and after the protocol amendment received CREN intravenously (IV).
- PCP PL - OLE CREN IV: Participants who on their PCP/parent study received placebo and who on this OLE study received CREN IV.
- PCP CREN SC - OLE CREN SC - OLE CREN IV: Participants who on their PCP/parent study received CREN and who on this OLE study initially received CREN SC and after the protocol amendment received CREN IV.
- PCP CREN IV - OLE CREN IV: Participants who on their PCP/parent study received CREN IV and who on this OLE study received CREN IV.
Period: Overall Study
Arm/Group | PCP PL - OLE CREN SC - OLE CREN IV | PCP PL - OLE CREN IV | PCP CREN SC - OLE CREN SC - OLE CREN IV | PCP CREN IV - OLE CREN IV
Started | 47 | 63 | 101 | 149
Completed | 20 | 27 | 44 | 59
Not Completed | 27 | 36 | 57 | 90
Not completed — Adverse Event | 4 | 1 | 4 | 5
Not completed — Death according to AE eCRF | 2 | 3 | 3 | 7
Not completed — Lost to Follow-up | 1 | 3 | 1 | 1
Not completed — Non-compliance | 0 | 1 | 3 | 3
Not completed — Non-compliance With Study Drug | 0 | 1 | 0 | 0
Not completed — Other Reason | 8 | 6 | 12 | 14
Not completed — Physician Decision | 1 | 3 | 4 | 11
Not completed — Protocol Violation | 1 | 1 | 3 | 1
Not completed — Withdrawal by Subject | 10 | 17 | 27 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCP PL - OLE CREN SC - OLE CREN IV | PCP PL - OLE CREN IV | PCP CREN SC - OLE CREN SC - OLE CREN IV | PCP CREN IV - OLE CREN IV | Total
Number analyzed (Participants) | 47 | 63 | 101 | 149 | 360
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.9 (7.4) | 71.9 (7.4) | 72.3 (7.2) | 72.2 (6.7) | 72.0 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 36 | 58 | 79 | 199
  Male | 21 | 27 | 43 | 70 | 161
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 4 | 10
  Not Hispanic or Latino | 45 | 61 | 98 | 145 | 349
  Not Stated | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 4 | 4
  Black or African American | 0 | 0 | 4 | 1 | 5
  White | 47 | 63 | 97 | 144 | 351

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. . An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to 50 months
Population: Safety Analysis population included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- PCP CREN - OLE CREN SC -OLE CREN IV: Participants who on their PCP/parent study received CREN and who on this OLE study initially received CREN SC and after the protocol amendment received CREN IV.
- PCP CREN - OLE CREN IV: Participants who on their PCP/parent study received CREN IV and who on this OLE study received CREN IV.
Arm/Group | PCP PL - OLE CREN SC - OLE CREN IV | PCP PL - OLE CREN IV | PCP CREN - OLE CREN SC -OLE CREN IV | PCP CREN - OLE CREN IV
Number analyzed (Participants) | 47 | 63 | 101 | 149
percentage of participants | 89.4 | 90.5 | 96.0 | 87.9

2. Primary Outcome: Percentage of Participants by Nature of AEs
Description: A serious adverse event (SAE) is any AE that meets any of the following criteria: fatal, life threatening, requires or prolongs inpatient hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect in a neonate/infant. Non-SAE of special interest for this study include the following: cerebral vascular edema, Superficial siderosis of central nervous system, cerebral micro-hemorrhages or macro-hemorrhages, pneumonia, liver injury.
Time Frame: Up to 50 months
Population: Safety Analysis population included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | PCP PL - OLE CREN SC - OLE CREN IV | PCP PL - OLE CREN IV | PCP CREN - OLE CREN SC -OLE CREN IV | PCP CREN - OLE CREN IV
Number analyzed (Participants) | 47 | 63 | 101 | 149
percentage of participants
  SAE | 19.1 | 22.2 | 21.8 | 23.5
  Non-SAE | 87.2 | 88.9 | 94.1 | 87.2

3. Primary Outcome: Percentage of Participants by Severity of AEs
Description: AE severity grading scale for the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0 was used for assessing adverse event severity. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on the following general guideline: Grade 1) mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, Grade 2) moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL), Grade 3) severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL, Grade 4) life-threatening consequences; urgent intervention indicated, Grade 5) death related to AE.
Time Frame: Up to 50 months
Population: Safety Analysis population included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | PCP PL - OLE CREN SC - OLE CREN IV | PCP PL - OLE CREN IV | PCP CREN - OLE CREN SC -OLE CREN IV | PCP CREN - OLE CREN IV
Number analyzed (Participants) | 47 | 63 | 101 | 149
percentage of participants
  Grade 1 | 19.1 | 34.9 | 29.7 | 22.1
  Grade 2 | 44.7 | 31.7 | 43.6 | 40.3
  Grade 3 | 12.8 | 17.5 | 16.8 | 19.5
  Grade 4 | 8.5 | 1.6 | 3.0 | 1.3
  Grade 5 | 4.3 | 4.8 | 3.0 | 4.7

4. Primary Outcome: Percentage of Participants With Human Anti-Therapeutic Antibody (ATA) Formation
Description: ATA is a measurement to explore the potential relationship of immunogenicity response with pharmacokinetics, safety and efficacy. Percentage of participants at post-baseline with positive results for ATA against crenezumab are reported.
Time Frame: Pre-dose (Day-14), predose at Week 25, 49, 97, Follow-up Week 8 (Week 153) and 12 (Week 157)
Population: Safety Analysis population included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | PCP PL - OLE CREN SC - OLE CREN IV | PCP PL - OLE CREN IV | PCP CREN - OLE CREN SC -OLE CREN IV | PCP CREN - OLE CREN IV
Number analyzed (Participants) | 47 | 63 | 101 | 149
percentage of participants | 9.1 | 3.4 | 9.1 | 0.7

5. Primary Outcome: Percentage of Participants With Amyloid-Related Imaging Abnormalities Edema/Effusions (ARIA-E)
Description: Alzheimer's disease (AD) is associated with ARIA. The occurrence of imaging abnormalities believed to represent cerebral vasogenic edema, has been reported in association with the investigational use of compounds that are intended to treat Alzheimer's disease by reducing Abeta in the brain. Here, the percentage of participants with symptomatic and asymptomatic ARIA-E were reported.
Time Frame: Baseline, Weeks 23, 47, 71, 97, 121 and 153
Population: Safety Analysis population included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | PCP PL - OLE CREN SC - OLE CREN IV | PCP PL - OLE CREN IV | PCP CREN - OLE CREN SC -OLE CREN IV | PCP CREN - OLE CREN IV
Number analyzed (Participants) | 47 | 63 | 101 | 149
percentage of participants
  Symptomatic | 0 | 0 | 0 | 0
  Asymptomatic | 0 | 0 | 0 | 0.7

6. Primary Outcome: Percentage of Participants With Amyloid-Related Imaging Abnormalities-Hemorrhage (ARIA-H)
Description: AD is associated with ARIA. Cerebral micro-hemorrhages (microbleeds [MBs]) are radiologically defined as small dot-like foci of signal loss observed on magnetic resonance imaging (MRI) sequences sensitive for paramagnetic tissue properties. The occurrence of MBs has also been identified as an adverse event in anti-amyloid vaccination trials, and together with superficial siderosis, they have been termed ARIA-H.
Time Frame: Baseline, Weeks 23, 47, 71, 97, 121 and 153
Population: Safety Analysis population included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | PCP PL - OLE CREN SC - OLE CREN IV | PCP PL - OLE CREN IV | PCP CREN - OLE CREN SC -OLE CREN IV | PCP CREN - OLE CREN IV
Number analyzed (Participants) | 47 | 63 | 101 | 149
percentage of participants
  Superficial Siderosis | 2.1 | 0 | 3.0 | 0.7
  New Micro-hemorrhage | 6.4 | 9.5 | 4.0 | 6.0

ADVERSE EVENTS:
Time Frame: Up to 50 months
Description: Safety Analysis population included all participants who received at least one dose of study drug.
Arm/Group | PCP PL - OLE CREN SC - OLE CREN IV | PCP PL - OLE CREN IV | PCP CREN SC - OLE CREN SC - OLE CREN IV | PCP CREN IV - OLE CREN IV
All-Cause Mortality (participants affected / at risk) | 2/47 | 3/63 | 3/101 | 7/149
Serious Adverse Events (participants affected / at risk) | 9/47 | 14/63 | 22/101 | 35/149
Other Adverse Events (participants affected / at risk) | 37/47 | 51/63 | 80/101 | 97/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCP PL - OLE CREN SC - OLE CREN IV (N=47) | PCP PL - OLE CREN IV (N=63) | PCP CREN SC - OLE CREN SC - OLE CREN IV (N=101) | PCP CREN IV - OLE CREN IV (N=149)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INCARCERATED HERNIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (5)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA ESCHERICHIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ADULT FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BASILAR ARTERY STENOSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEMENTIA (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
DEMENTIA WITH LEWY BODIES (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EPILEPSY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
SYNCOPE (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DEVICE DISLOCATION (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEVICE FAILURE (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AGGRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
DISORIENTATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PULMONARY GRANULOMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AORTIC ANEURYSM (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
EXSANGUINATION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCP PL - OLE CREN SC - OLE CREN IV (N=47) | PCP PL - OLE CREN IV (N=63) | PCP CREN SC - OLE CREN SC - OLE CREN IV (N=101) | PCP CREN IV - OLE CREN IV (N=149)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3) | 5 (5)
DIARRHOEA (Gastrointestinal disorders) | 6 (7) | 3 (3) | 11 (12) | 14 (23)
VOMITING (Gastrointestinal disorders) | 0 (0) | 3 (5) | 5 (6) | 8 (11)
FATIGUE (General disorders) | 2 (2) | 0 (0) | 8 (8) | 4 (4)
INJECTION SITE ERYTHEMA (General disorders) | 2 (13) | 1 (1) | 8 (10) | 2 (2)
INJECTION SITE EXTRAVASATION (General disorders) | 3 (5) | 1 (1) | 3 (7) | 4 (16)
BRONCHITIS (Infections and infestations) | 2 (2) | 2 (2) | 4 (5) | 9 (9)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (7) | 5 (5) | 15 (20) | 13 (15)
URINARY TRACT INFECTION (Infections and infestations) | 7 (8) | 9 (13) | 16 (23) | 18 (34)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (7) | 11 (14) | 10 (11) | 13 (13)
CONTUSION (Injury, poisoning and procedural complications) | 2 (6) | 2 (2) | 6 (8) | 8 (10)
FALL (Injury, poisoning and procedural complications) | 7 (10) | 8 (11) | 26 (42) | 18 (28)
LACERATION (Injury, poisoning and procedural complications) | 3 (3) | 2 (3) | 10 (11) | 7 (7)
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 5 (5) | 3 (5)
WEIGHT DECREASED (Investigations) | 4 (4) | 2 (2) | 8 (11) | 7 (7)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (4) | 5 (6) | 8 (10) | 8 (10)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5) | 7 (7) | 8 (8)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 4 (6) | 1 (2)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (8) | 1 (1) | 2 (2) | 0 (0)
CEREBRAL MICROHAEMORRHAGE (Nervous system disorders) | 3 (3) | 4 (5) | 3 (3) | 6 (7)
DIZZINESS (Nervous system disorders) | 2 (2) | 5 (5) | 11 (14) | 10 (11)
HEADACHE (Nervous system disorders) | 1 (1) | 2 (2) | 8 (10) | 3 (4)
AGITATION (Psychiatric disorders) | 9 (9) | 4 (4) | 13 (20) | 13 (14)
ANXIETY (Psychiatric disorders) | 1 (1) | 4 (4) | 8 (9) | 15 (16)
CONFUSIONAL STATE (Psychiatric disorders) | 3 (3) | 1 (1) | 3 (4) | 3 (4)
DELUSION (Psychiatric disorders) | 3 (3) | 1 (1) | 7 (7) | 4 (6)
DEPRESSION (Psychiatric disorders) | 3 (3) | 8 (9) | 5 (5) | 7 (7)
INSOMNIA (Psychiatric disorders) | 3 (6) | 1 (1) | 8 (10) | 8 (9)
URINARY INCONTINENCE (Renal and urinary disorders) | 4 (4) | 0 (0) | 5 (6) | 8 (8)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (11) | 3 (3) | 8 (9) | 11 (13)
RASH (Skin and subcutaneous tissue disorders) | 2 (7) | 5 (5) | 2 (2) | 6 (7)
HAEMATOMA (Vascular disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT01723826/Prot_SAP_000.pdf